CLINICAL TRIAL: NCT00498940
Title: Biventricular Pacing After Cardiopulmonary Bypass
Acronym: BIPACS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Accrual too slow; grant renewal unlikely; AAI as effective as BiV in Phase III
Sponsor: Henry M. Spotnitz (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Henry M. Spotnitz, George H. Humphreys, II Professor of Surgery, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAB5600; R01HL080152 (NIH)
Record Dates: First submitted 2007-07-09; First posted 2007-07-11 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure
Keywords: LV function, Compliance, wall motion, echocardiography
MeSH Terms: conditions — Heart Failure; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Biventricular Pacing (Active Comparator): After weaning from bypass, patients received temporary biventricular pacing for 24 hours. Values obtained from optimization testing determined pacemaker settings (AVD, VVD, heart rate).
  Interventions: Device: Optimization Testing; Device: Temporary Biventricular Pacing
- Standard of Care (Active Comparator): No continuous pacing occurred about surgery. Patients underwent optimization testing.
  Interventions: Device: Optimization Testing

INTERVENTIONS:
Device: Optimization Testing — Atrioventricular (AVD) and interventricular (VVD) delays and left ventricle lead site location were optimized after weaning off bypass (Phase I), after sternal closure (Phase II), and 12 to 24 hours (Phase III) after bypass. Intrinsic heart rate was also optimized in Phase III.
  Other Names: Medtronic Insync III
Device: Temporary Biventricular Pacing — Continuous temporary biventricular pacing for 24 hours at a heart rate of 90 bpm or 10 bpm above intrinsic heart rate.
  Arms: Biventricular Pacing

SUMMARY:
The purpose of this study is to investigate the efficacy of optimized temporary biventricular pacing (BiVP) in patients undergoing open-heart surgery with preoperative LV dysfunction and an intraventricular conduction delay. This study will compare extended temporary biventricular pacing versus standard of care by assessing patients randomized to the two groups, from the conclusion of cardiopulmonary bypass, until the conclusion of pharmacologic circulatory support in the intensive care unit. In addition, effects of biventricular pacing will be tested in all patients, at three time points, using different measures of blood flow. Results from this research will demonstrate whether temporary BiVP improves cardiac output after open-heart surgery and whether ventricular pacing optimization increases cardiac output in this setting. Success would lead to the development of recommendations for use of BiVP postoperatively and would stimulate the development of pacemakers with appropriate features.

The primary hypothesis is that the optimum pacing protocol (POPT) will increase cardiac index (CI) by 15% (from approximately 2.30 to 2.64 L/min/m2) compared to standard of care as measured by thermodilution 12-24 hours postoperatively. Secondary objectives include defining POPT at three time points within 24 hours of surgery. The investigator will examine which forms of cardiac dysfunction benefit from temporary pacing using direct and indirect measures of perfusion and cardiac function. The investigator will also analyze survival, length of stay, incidence of arrhythmias, and cost of postoperative care.

DETAILED DESCRIPTION:
Biventricular pacing (BiVP) reverses intraventricular conduction delay (IVCD) and left ventricular (LV) dysfunction in dilated cardiomyopathy (DCM). BiVP improves LV function and cardiac index (Cl) at no energy cost. In the MIRACLE trial, in patients with DCM, IVCD and LV ejection fraction <35%, demonstrated improved subjective and objective measures of exercise tolerance and cardiac function with BiVP. BiVP benefits many, but selection criteria are not fully developed, and 30% of recipients are "nonresponders," at a cost of more than $2 billion/year. Preliminary data suggest that BiVP can benefit patients with low output states after cardiac surgery. This study will assess surgical application of BiVP while assessing mechanisms of action and optimization. 190 cardiac surgery patients will be randomized with LV dysfunction preoperatively to paced and standard of care groups. BiVP will be optimized and continued postoperatively until patients are stable. BiVP will be assessed transiently in all patients at three time points. The primary end point is a 15% improvement in thermal dilution Cl measured in the intensive care unit (ICU). Effects of heart rate, atrioventricular delay, ventricular pacing site, and interventricular delay on Cl will be assessed using a randomized sequence of data collection. Secondary endpoints include incidence of arrhythmias, inotropic support, urine output, weight gain, morbidity, mortality, and ICU costs. These studies are important because of a high probability of clinical benefit. The methods employed will provide precision, breadth of measurement, and range of pacing sites superior to any other setting. The protocol will provide new and important scientific information that will benefit not only surgical patients but also the general population of BiVP recipients.

ELIGIBILITY:
Inclusion Criteria:

* LV ejection fraction < 41%
* QRS duration > 99 msec

Or:

* Mitral and Aortic Valve Repair or Replacement

Exclusion Criteria:

* Congenital Heart Disease
* Intracardiac Shunts
* Preoperative Pacing for Heart Block (2nd or 3rd degree) or Sinus Bradycardia
* Heart Rate > 120 beats per min after Cardiopulmonary Bypass
* Preoperative Atrial Fibrillation
* Previous Cardiac Surgery
* Inability to undergo biventricular pacing prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry M. Spotnitz, M.D., Principal Investigator — Professor
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Rubinstein BJ, Wang DY, Cabreriza SE, Cheng B, Aponte-Patel L, Murata A, Rusanov A, Richmond ME, Quinn TA, Spotnitz HM. Response of mean arterial pressure to temporary biventricular pacing after chest closure during cardiac surgery. J Thorac Cardiovasc Surg. 2012 Dec;144(6):1445-52. doi: 10.1016/j.jtcvs.2012.04.026. Epub 2012 Aug 21. PMID 22920599
- See also: ColumbiaDoctors - Clinical Trials Search Tool — http://sklad.cumc.columbia.edu/surgery/clinicaltrials/View_Trial.php?ID=9

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began on April 1, 2007 and ended March 1, 2012. The trial was conducted at Columbia University and University of California, Lost Angeles.
Pre-assignment Details: Enrolled patients not meeting study criteria just prior to the start of study, withdrawn at surgeon's discretion, or change in surgery type were not randomized. 61 out of the 111 enrolled subjects were randomized, received study intervention and had data analyzed.
Groups:
- Biventricular Pacing: After weaning from bypass, patients will receive temporary biventricular pacing for 24 hours. Values obtained from optimization testing will determine pacemaker settings (AVD, VVD, heart rate).
  Optimization Testing: Atrioventricular (AVD) and interventricular (VVD) delays and heart rate were optimized after weaning off bypass (phase I), after sternal closure (phase II), and 12 to 24 hours (phase III) after bypass.
  Temporary Biventricular Pacing: Continuous temporary biventricular pacing for 24 hours.
- Standard of Care: No post operative pacing is to occur. Patients will undergo optimization testing.
  Optimization Testing: Atrioventricular (AVD) and interventricular (VVD) delays and heart rate were optimized after weaning off bypass (phase I), after sternal closure (phase II), and 12 to 24 hours (phase III) after bypass.
Period: Overall Study
Arm/Group | Biventricular Pacing | Standard of Care
Started | 30 | 31
Completed | 30 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biventricular Pacing | Standard of Care | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (11.2) | 67.9 (11.7) | 67.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 21 | 24 | 45
Ejection Fraction (%) [Mean (Standard Deviation); unit: percentage of ventricular blood pumped] | 34 (.1) | 32 (.2) | 33 (.1)
QRS duration (ms) [Mean (Standard Deviation); unit: msec] | 120.1 (27.9) | 118.6 (23.0) | 119.3 (25.3)

OUTCOME MEASURES:

1. Primary Outcome: Thermal Dilution Cardiac Index (CI) Measured in the Intensive Care Unit (ICU).
Description: Cardiac output (CO) 12-24 hours after bypass is measured five times and averaged. CO is then converted to CI, after division by the patient's body surface area.
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: L/min/m^2
Arm/Group | Biventricular Pacing | Standard of Care
Number analyzed (Participants) | 23 | 24
L/min/m^2 | 2.83 (.16) | 2.52 (.13)
Statistical Analysis 1: Comparison: Biventricular Pacing vs Standard of Care; Test type: Superiority or Other; p = .14, t-test, 2 sided — Differences in cardiac index between groups were assessed by an independent 2-sample t test

2. Secondary Outcome: Number of Subjects With Postoperative Complications
Description: This is to measure the total number of subjects that experienced any of the following complications: sepsis/infection, renal failure, respiratory failure/complications, bleeding requiring reoperation, cerebrovascular accident.
Time Frame: 30 days after surgery
Measure: Number; unit: participants
Arm/Group | Biventricular Pacing | Standard of Care
Number analyzed (Participants) | 30 | 31
participants | 10 | 10

ADVERSE EVENTS:
Arm/Group | Biventricular Pacing | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 1/30 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biventricular Pacing (N=30) | Standard of Care (N=31)
Bleeding at lead site (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No